CLINICAL TRIAL: NCT00858702
Title: Add-on Study of CCBs or Diuretics in Essential Hypertension Not Achieving Target Blood Pressure on Olmesartan Medoxomil Alone
Brief Title: Calcium Channel Blockers (CCBs) or Diuretics as an Add-on to Olmesartan Medoxomil in Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Yoshihiro Kakehi, Daiichi Sankyo Co., Ltd.
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OLM004-071
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
Keywords: Essential hypertension; Combination therapy
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): olmesartan medoxomil tablets and a CCB tablet (of the dihydropyridine class), once daily for 8 weeks
  Interventions: Drug: olmesartan medoxomil and a CCB
- 2 (Experimental): olmesartan medoxomil and a diuretic tablet (of the thiazide class)
  Interventions: Drug: olmesartan medoxomil and a diuretic

INTERVENTIONS:
Drug: olmesartan medoxomil and a CCB — olmesartan medoxomil tablets and a CCB tablet once daily for 8 weeks
  Arms: 1
Drug: olmesartan medoxomil and a diuretic — olmesartan medoxomil tablets and a diuretic tablet, once daily for 8 weeks
  Arms: 2

SUMMARY:
The purpose of the study is to test the efficacy and safety of the combination of Calcium Channel Blockers (CCBs)(of the dihydropyridine class) or Diuretics (of the thiazide class) and olmesartan medoxomil in essential hypertensive patients whose blood pressure is not adequately controlled with olmesartan medoxomil alone

ELIGIBILITY:
Inclusion Criteria:

* Mean seated blood pressure greater than or equal to 140/90 mmHg under circumstances in pre-treatment with olmesartan medoxomil
* Mean 24-hour blood pressure evaluated by ambulatory blood pressure monitoring greater than or equal to 135/80 mmHg under circumstances in pre-treatment with olmesartan medoxomil

Exclusion Criteria:

* Patients with secondary hypertension
* Any serious disorder which may limit the ability to evaluate the efficacy or safety of the test drugs

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-02; Primary Completion 2005-07 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Research and Development Division, Study Director — Daiichi Sankyo Co., Ltd.
Locations (1):
- Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 172 patients were enrolled at 5 centers in Japan from February 12, 2005 to April 30, 2005.
Pre-assignment Details: After the 4 to 6 weeks of olmesartan medoxomil monotherapy period, 105 patients who met the entry criteria for the combination therapy period were randomized to calcium channel blocker (of the dihydropyridine class) combination group or diuretic (of the thiazide class)combination group.
Groups:
- Olmesartan Tablets and a Calcium Channel Blocker Tablet: olmesartan medoxomil tablets and a calcium channel blocker tablet (of the dihydropyridine class), once daily for 8 weeks
- Olmesartan Medoxomil Tablets and a Diuretic Tablet: olmesartan medoxomil tablets and a diuretic tablet (of the thiazide class)once daily for 8 weeks
Period: Overall Study
Arm/Group | Olmesartan Tablets and a Calcium Channel Blocker Tablet | Olmesartan Medoxomil Tablets and a Diuretic Tablet
Started | 53 | 52
Completed | 48 | 50
Not Completed | 5 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Other | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Olmesartan Tablets and a Calcium Channel Blocker Tablet: olmesartan medoxomil tablets and a calcium channel blocker tablet, once daily for 8 weeks
- Olmesartan Medoxomil Tablets and a Diuretic: olmesartan medoxomil tablets and a diuretic once daily for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Olmesartan Tablets and a Calcium Channel Blocker Tablet | Olmesartan Medoxomil Tablets and a Diuretic | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.2) | 57.4 (9.4) | 56.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 31 | 32 | 63
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 53 | 52 | 105
Region of Enrollment [Number; unit: participants]
  Japan | 53 | 52 | 105

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Achieving Target Sitting Blood Pressure of Less Than 130/85
Time Frame: Baseline to week 8
Population: Primary analysis was conducted for full analysis set. It excluded the patients who were not administrated study drugs, or did not satisfy entry criteria, or had no data after randomisation.
Measure: Number; unit: Percent of participants
Groups:
- Olmesartan Medoxomil Tablets and a Diuretic: olmesartan medoxomil tablets and a diuretic tablet (of the thiazide class) once daily for 8 weeks
Arm/Group | Olmesartan Tablets and a Calcium Channel Blocker Tablet | Olmesartan Medoxomil Tablets and a Diuretic
Number analyzed (Participants) | 50 | 49
Percent of participants | 34.0 | 59.2
Statistical Analysis 1: Comparison: Olmesartan Tablets and a Calcium Channel Blocker Tablet vs Olmesartan Medoxomil Tablets and a Diuretic; Test type: Superiority or Other; p = 0.0158, Fisher Exact — No consideration for multiplicity

2. Secondary Outcome: Percentage of Patients With Drug-related Adverse Events (Subjective Symptoms/Objective Findings)
Description: Drug-related adverse events are adverse events(AEs) as determined by the Investigator that can not be denied to be related to the study drugs. The relationship between adverse events and drugs were determined by the Investigator based on his/her clinical judgement. Factors used in determining relatedness included, but are not limited to, the medical history of the participant, use of concomitant medication, and the time course from drug administration to AE occurence.
Time Frame: At week 8
Population: Safety analysis (Clinical AEs:subjective symptoms / objective findings) was conducted for Safety Population. It excluded the patients who were not administrated study drugs.
Measure: Number; unit: Percent of participants
Groups:
- Olmesartan Tablets and a Calcium Channel Blocker Tablet: olmesartan medoxomil tablets and a calcium channel blocker (of the dihydropyridine class) tablet, once daily for 8 weeks
Arm/Group | Olmesartan Tablets and a Calcium Channel Blocker Tablet | Olmesartan Medoxomil Tablets and a Diuretic
Number analyzed (Participants) | 53 | 52
Percent of participants | 0 | 7.7
Statistical Analysis 1: Comparison: Olmesartan Tablets and a Calcium Channel Blocker Tablet vs Olmesartan Medoxomil Tablets and a Diuretic; Test type: Superiority or Other; p = 0.0566, Fisher Exact — No consideration for multiplicity

3. Secondary Outcome: Percent of Patients With Drug-related Adverse Events (Laboratory Changes in Clinical Laboratory Values)
Description: Drug-related, laboratory value change adverse events are adverse events(AEs) as determined by the Investigator that can not be denied to be related to the study drugs. The relationship between adverse events and drugs were determined by the Investigator based on his/her clinical judgement. Factors used in determining relatedness included, but are not limited to, the medical history of the participant, use of concomitant medication, and the time course from drug administration to AE occurence.
Time Frame: At week 8
Population: Safety analysis (laboratory AEs:abnormal changes in clinical laboratory values) was conducted for Safety Population. It excluded the patients who were not administered study drugs, or had no clinical laboratory data.
Measure: Number; unit: Percent of participants
Groups:
- Olmesartan Medoxomil Tablets and a Diuretic: olmesartan medoxomil tablets and a diuretic tablet(of the the thiazide class) once daily for 8 weeks
Arm/Group | Olmesartan Tablets and a Calcium Channel Blocker Tablet | Olmesartan Medoxomil Tablets and a Diuretic
Number analyzed (Participants) | 52 | 52
Percent of participants | 1.9 | 44.2
Statistical Analysis 1: Comparison: Olmesartan Tablets and a Calcium Channel Blocker Tablet vs Olmesartan Medoxomil Tablets and a Diuretic; Test type: Superiority or Other; p < 0.001, Fisher Exact — No consideration for multiplicity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No